CLINICAL TRIAL: NCT02966782
Title: A Phase 1b Study Evaluating the Safety and Pharmacokinetics of Venetoclax as a Single-Agent and in Combination With Azacitidine in Subjects With Relapsed/Refractory Myelodysplastic Syndromes
Brief Title: A Study Evaluating Venetoclax Alone and in Combination With Azacitidine in Participants With Relapsed/Refractory Myelodysplastic Syndromes (MDS)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Collaborators: Celgene; Genentech, Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M15-522; 2016-001904-46 (EudraCT Number)
Record Dates: First submitted 2016-11-15; First posted 2016-11-17 (Estimated); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Myelodysplastic Syndromes (MDS)
Keywords: Relapsed/refractory; Venetoclax; Azacitidine
MeSH Terms: conditions — Myelodysplastic Syndromes; Recurrence | interventions — venetoclax; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Venetoclax monotherapy (Cohort 1) (Experimental)
  Interventions: Drug: venetoclax
- Venetoclax + azacitidine (Cohort 2) (Experimental)
  Interventions: Drug: venetoclax; Drug: azacitidine
- Safety Expansion (Cohort 3) (Experimental)
  Interventions: Drug: venetoclax; Drug: azacitidine

INTERVENTIONS:
Drug: venetoclax — Tablet
  Other Names: ABT-199; GDC-0199
Drug: azacitidine — Powder for injection, subcutaneously or intravenous
  Other Names: Vidaza
  Arms: Safety Expansion (Cohort 3); Venetoclax + azacitidine (Cohort 2)

SUMMARY:
This is a Phase 1b, open-label, multicenter study designed to evaluate the safety and pharmacokinetics of venetoclax as a single-agent and in combination with azacitidine in participants with relapsed/refractory Myelodysplastic Syndromes (MDS).

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have relapsed or refractory MDS.
* Subject enrolled in venetoclax monotherapy must have documented failure of prior therapy with a hypomethylating agent (HMA). HMA-failure is defined as:

  1. Relapse after initial complete or partial response or hematological improvement after at least 4 cycles of azacitidine or at least 4 cycles of decitabine within the last 5 years, OR
  2. Failure to achieve complete or partial response or hematological improvement after at least 4 cycles of azacitidine or at least 4 cycles of decitabine within the last 5 years
* Subjects must have presence of < 20% bone marrow blasts per bone marrow biopsy/aspirate at screening.
* Subject is not a candidate to undergo allogenic hematopoietic stem cell transplantation (HSCT).
* Subject must have an Eastern Cooperative Oncology Group (ECOG) performance score of ≤2.
* Subject must have adequate hematologic, renal, and hepatic function.

Exclusion Criteria:

* Subject has received prior therapy with a BH3 mimetic.
* Subject has MDS evolving from a pre-existing myeloproliferative neoplasm (MPN).
* Subject has MDS/MPN including chronic myelomonocytic leukemia (CMML), atypical chronic myeloid leukemia (CML), juvenile myelomonocytic leukemia (JMML) and unclassifiable MDS/MPN.
* Subject has received allogeneic HSCT or solid organ transplantation.
* Subject has received a live attenuated vaccine within 4 weeks prior to the first dose of study drug.
* Subject is pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2017-03-07 (Actual); Primary Completion 2023-04-05 (Actual); Study Completion 2023-04-05 (Actual)

PRIMARY OUTCOMES:
AUCt for azacitidine | Up to 32 days
  Area under the plasma concentration-time curve (AUC) from 0 to the time of the last measurable concentration (AUCt) for azacitidine
Clearance (CL) for azacitidine | Up to 32 days
Cmax for azacitidine | Up to 32 days
  Maximum plasma concentration (Cmax) of azacitidine
Tmax for venetoclax | Up to 32 days
  Time to Cmax (peak time, Tmax) for venetoclax
Recommended Phase 2 Dose (RPTD) and dosing schedules of venetoclax as monotherapy and in combination with azacitidine | Measured from Day 1 until day 28 per dose level.
AUC[0 to infinity] for azacitidine | Up to 32 days
  Area under the plasma concentration-time curve from Time 0 to infinite time.
Tmax for azacitidine | Up to 32 days
  Time to Cmax (peak time, Tmax) for azacitidine
AUC [0-24] for venetoclax | Up to 32 days
  AUC over a 24-hour dose interval (AUC[0-24]) for venetoclax
AUCt for venetoclax | Up to 32 days
  Area under the plasma concentration-time curve (AUC) from 0 to the time of the last measurable concentration (AUCt) for venetoclax
Cmax of venetoclax | Up to 32 days
  Maximum plasma concentration (Cmax) of venetoclax
Half-life (t[1/2]) for azacitidine | Up to 32 days
  Terminal elimination half-life (t[1/2]) for azacitidine
Number of Participants With Adverse Events (AEs) | Up to Maximum of 24 months
  An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment. The investigator assesses the relationship of each event to the use of study. A serious adverse event (SAE) is an event that results in death, is life-threatening, requires or prolongs hospitalization, results in a congenital anomaly, persistent or significant disability/incapacity or is an important medical event that, based on medical judgment, may jeopardize the participant and may require medical or surgical intervention to prevent any of the outcomes listed above. Treatment-emergent adverse events/treatment-emergent serious adverse events (TEAEs/TESAEs) are defined as any event that began or worsened in severity on or after the first dose of study drug.

SECONDARY OUTCOMES:
Event-Free Survival (EFS) | Measured from the date of the first dose of study drug to date of earliest disease progression, death, or initiation of new non-protocol-specified anti-MDS therapy without documented progression, and for up to 5 years after the last subject is enrolled.
Overall Survival (OS) | Measured from the date of first dose of study drug to the date of death, and for up to 5 years after the last subject is enrolled.
Rate of Modified Overall Response (mORR) | Measured from Cycle 1 Day 1 (C1D1) as long as the subject continues to benefit, or until the occurrence of unacceptable toxicity, death, exercise of investigator discretion, or withdrawal of consent, and for an anticipated maximum duration of 24 months.
  Proportion of participants with a mORR using best outcome will be calculated.
Time to next treatment (TTNT) | Measured from first dose of study drug to start of new non-protocol specified MDS therapy, and for up to 5 years after the last subject is enrolled.
Duration of mORR | Measured from the date of first response (CR, mCR or PR) to the earliest documentation of progressive disease (PD), and for an anticipated maximum duration of 24 months.
  Defined as the number of days from the date of first response (CR, mCR or PR) to the earliest documentation of progressive disease or death of any cause, whichever occurs earlier..
Rate of platelet (PLT) transfusion independence | Measured from Cycle 1 Day 1 as long as the subject continues to benefit, or until the occurrence of unacceptable toxicity, death, exercise of investigator discretion, or withdrawal of consent, and for an anticipated maximum duration of 24 months.
  Proportion of participants who become platelet transfusion-independent
Time to Transformation acute myeloid leukemia (AML) | Measured from the date of first dose of study drug to the date of documented AML transformation for an anticipated maximum duration of 24 months.
  Defined as blast count greater than or equal to 20% in either peripheral blood or bone marrow.
Progression-Free Survival (PFS) | Measured from the date of the first dose of study drug to the date of earliest disease progression or death, and for an anticipated maximum duration of 24 months.
Overall Response Rate (ORR) | Measured from Cycle 1 Day 1 as long as the subject continues to benefit, or until the occurrence of unacceptable toxicity, death, exercise of investigator discretion, or withdrawal of consent, and for an anticipated maximum duration of 24 months.
  ORR (equals the sum of rates of complete remission [CR] + marrow complete remission (mCR) + partial remission [PR]) of venetoclax as a single-agent and in combination with azacitidine.
Complete Remission (CR) Rate | Measured from Cycle 1 Day 1 as long as the subject continues to benefit, or until the occurrence of unacceptable toxicity, death, exercise of investigator discretion, or withdrawal of consent, and for an anticipated maximum duration of 24 months.
  Proportion of subjects who achieved a complete remission.
Rate of red blood cell (RBC) transfusion independence | Measured from Cycle 1 Day 1 as long as the subject continues to benefit, or until the occurrence of unacceptable toxicity, death, exercise of investigator discretion, or withdrawal of consent, and for an anticipated maximum duration of 24 months.
  Proportion of red blood cell (RBC) transfusion independence.
Duration of Complete Response (CR) | Measured from date of first response (CR) to the to the earliest documentation of progressive disease or death of any cause, and for an anticipated maximum duration of 24 months.
  Duration of CR will be defined as the number of days from the date of first response CR to the earliest documentation of progressive disease or death of any cause, whichever occurs earlier.
Rate of Hematologic Improvement (HI) | Measured from Cycle 1 Day 1 as long as the subject continues to benefit, or until the occurrence of unacceptable toxicity, death, exercise of investigator discretion, or withdrawal of consent, and for an anticipated maximum duration of 24 months.
  Proportion of participants with HI (erythroid/platelet/neutrophil responses)
Rate of marrow complete remission (mCR) | Measured from Cycle 1 Day 1 (C1D1) as long as the subject continues to benefit, or until the occurrence of unacceptable toxicity, death, exercise of investigator discretion, or withdrawal of consent, and for an anticipated maximum duration of 24 months.
  Proportion of participants with marrow complete remission with or without hematological improvement.
Duration of ORR | Measured from the date of first response (CR or PR) to the earliest documentation of progressive disease or death of any cause, and for an anticipated maximum duration of 24 months.
  Duration of response (ORR) will be defined as the number of days from the date of first response (CR or PR) to the earliest documentation of progressive disease or death of any cause, whichever occurs earlier.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (23):
- United States (10):
  - University of Arizona Cancer Center - North Campus /ID# 157503, Tucson, Arizona
  - University of Colorado Hospital /ID# 155365, Aurora, Colorado
  - Yale University /ID# 162544, New Haven, Connecticut
  - Duplicate_University of Chicago /ID# 155364, Chicago, Illinois
  - Pediatric Endocrine Associates /ID# 171227, Boston, Massachusetts
  - Dana-Farber Cancer Institute /ID# 155361, Boston, Massachusetts
  - University of Massachusetts - Worcester /ID# 155366, Worcester, Massachusetts
  - Columbia Univ Medical Center /ID# 156388, New York, New York
  - Oregon Health and Science University /ID# 155360, Portland, Oregon
  - University of Texas MD Anderson Cancer Center /ID# 155362, Houston, Texas
- Australia (5):
  - St George Hospital /ID# 156037, Kogarah, New South Wales
  - Liverpool Hospital /ID# 155952, Liverpool, New South Wales
  - St Vincent's Hospital Melbourne /ID# 155950, Fitzroy Melbourne, Victoria
  - The Royal Melbourne Hospital /ID# 155949, Parkville, Victoria
  - Royal Perth Hospital /ID# 155951, Perth, Western Australia
- Germany (8):
  - Universitatsklinikum Mannheim /ID# 156038, Mannheim, Baden-Wurttemberg
  - Universitaetsklinikum Koeln /ID# 155519, Cologne, North Rhine-Westphalia
  - Universitaetsklinikum Duesseldorf /ID# 154899, Düsseldorf, North Rhine-Westphalia
  - Marien Hospital Duesseldorf /ID# 155518, Düsseldorf, North Rhine-Westphalia
  - Universitaetsklinikum Leipzig /ID# 154897, Leipzig, Saxony
  - Universitaetsklinikum Carl Gustav Carus an der TU Dresden /ID# 154898, Dresden
  - Universitaetsklinikum Halle (Saale) /ID# 158643, Halle
  - Klinikum rechts der Isar - Technische Universitaet Muenchen /ID# 154896, Munich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zeidan AM, Borate U, Pollyea DA, Brunner AM, Roncolato F, Garcia JS, Filshie R, Odenike O, Watson AM, Krishnadasan R, Bajel A, Naqvi K, Zha J, Cheng WH, Zhou Y, Hoffman D, Harb JG, Potluri J, Garcia-Manero G. A phase 1b study of venetoclax and azacitidine combination in patients with relapsed or refractory myelodysplastic syndromes. Am J Hematol. 2023 Feb;98(2):272-281. doi: 10.1002/ajh.26771. Epub 2022 Nov 10. PMID 36309981
- [Derived] Franke GN, Luckemeier P, Platzbecker U. Allogeneic Stem-Cell Transplantation in Patients With Myelodysplastic Syndromes and Prevention of Relapse. Clin Lymphoma Myeloma Leuk. 2021 Jan;21(1):1-7. doi: 10.1016/j.clml.2020.10.008. Epub 2020 Oct 16. PMID 33191169